CLINICAL TRIAL: NCT04250285
Title: University of Bojnord
Brief Title: Academic Self-regulation, Parenting Dimensions and Academic Procrastination
Status: Completed | Type: Observational
Sponsor: Malahat Amani (Other)
Responsible Party: Sponsor-Investigator, Malahat Amani, assistant professor, University of Bojnord
Organization: University of Bojnord (Other)
Other Study IDs: 131709
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Self-regulation; Parenting; Procrastination
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive method — After obtaining relevant permissions from the university and organization of education and selecting participants, the study was explained for students and their satisfaction obtained. Then questionnaires were given to participants. To observe ethical considerations, questionnaires were anonymous and has been confided that the participants' responses was maintained in the study and is not given anyone
  Other Names: correlation

SUMMARY:
the method was the correlational way. The statistical population of the was all of the boy students of the second-period elementary school in Garmeh city (Iran). the sample size was 278. The age of participants was in the range of 9 to13 years old.

ELIGIBILITY:
Inclusion Criteria:

be the male student, having the age of 9 to 13 years, having the ability of reading and writing

Exclusion Criteria:

* be female, no be student, no having age of 9 to 13 years, disability of reading and writing, having psychotic disorders

Ages: 9 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — self-representation
Study Population: male students in age range of 9 to 13 years old in Garmeh city(Iran)
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Self-Regulation | 2 days
  self-regulation was measured by the Academic Self-Regulation Questionnaire. this questionnaire has 30 items to measure memory, targeting, self-evaluation, assistance, responsibility and organization strategies. items are assessed on a six-point score of never (1), rarely (2), sometimes (3), usually (4), most times (5) and always (6). the high scores indicate level high of the self regulation
Procrastination | 2 days
  procrastination was measured by Procrastination Academic Scale. This scale has 27 items that examine components of preparation for exams, preparation for tasks and preparation class projects. It is responded to items on a four-point scale namely, "rarely", "sometimes", "most" and "always".the high scores indicate the high level of procrastination.
parenting | 2 days
  parenting was measured by the Scale of parenting style. This scale has parental responsiveness and parental control dimension. Items measure the adolescents' perception from their parents' responsiveness and control. The scale of parenting style has 38 items and it is responded on the five-point scale as "always true" to "always false". the high scores indicated the high level in control and responsiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Malahat Amani, Bojnourd, North Khorasan, Iran

IPD SHARING:
Plan to Share IPD: No